CLINICAL TRIAL: NCT07357207
Title: Video-immunotherapy: a New Approach in Breast Cancer Treatment
Acronym: VIT-BC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Biomedicine and Genome Center (Other Government)
Collaborators: Antalya Training and Research Hospital (Other Government); Akdeniz University Hospital (Other); Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Duygu Sag, Assoc. Prof., Izmir Biomedicine and Genome Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: iBG-2022-017; 121C245 (Other Grant/Funding Number: Scientific And Technological Research Council of Turkey)
Record Dates: First submitted 2025-11-27; First posted 2026-01-21 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Female Breast Cancer Patients
Keywords: video-immunotherapy

STUDY DESIGN:
Intervention Model Description: In this study, locally advanced breast cancer patients who received neoadjuvant chemotherapy as routine treatment for 5-6 months will be randomized into 2 groups: EXPERIMENT GROUP: will play the "video-immunotherapy" about immune cells fighting breast cancer (n=40). CONTROL GROUP: Will play the placebo video game (n=40). The study will be terminated at the end of 5-6 months when the patients undergo surgery as a normal treatment process.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video-immunotherapy group (Experimental): EXPERIMENT GROUP: will play the "video-immunotherapy" about immune cells fighting breast cancer.
  Interventions: Behavioral: UMAY - Video-immunotherapy game
- Control group (Placebo Comparator): CONTROL GROUP: the placebo video game.
  Interventions: Behavioral: Control - Plasebo Game

INTERVENTIONS:
Behavioral: UMAY - Video-immunotherapy game — "UMAY" video-immunotherapy about immune cells fighting breast cancer - participants will play the UMAY video game offered as a mobile phone app at home for at least 20 minutes at least 4 days a week.
  Arms: Video-immunotherapy group
Behavioral: Control - Plasebo Game — participants will play the placebo video game as a mobile phone app at home for at least 20 minutes at least 4 days a week.
  Arms: Control group

SUMMARY:
Breast cancer is the most common type of cancer among women worldwide and in Türkiye and remains one of the leading causes of cancer-related mortality. The high mortality rate and the fact that the disease severely reduces patients' quality of life create an urgent need for the development of innovative therapeutic approaches. Cancer immunotherapy aims to inhibit tumor growth and spread by harnessing the immune system. The fact that the immune system interacts with the nervous system and the endocrine system reveals that the integrity of the body and mind is very important in strengthening the immune system against cancer. Within the scope of psychoneuroimmunology, studies such as meditation, breathing therapy, hypnosis, and yoga have an indirect effect on the immune system by reducing the stress level of the person and improving the psychology, while techniques such as guided imagery can play a direct role in regulating the immune system. It has been shown that guided imagery studies, which can create unexpected effects thanks to the inability of the human mind to distinguish between imagination and reality, can increase the activity of immune cells with anti-tumoral activity in cancer patients and even reduce patient mortality. In addition to the cytotoxic activities of immune system cells, imagery can also have an effect on the regulation of tissue migration. Therefore, guided imagery studies in breast cancer patients can contribute both to immune system regulation and to increase lymphocyte migration to the tumor tissue of patients if they are applied effectively and long-term enough. In guided imagery studies, it is thought that the effectiveness is limited by the stress experienced by the patients/subjects during the effort of practicing imagery. In addition, imagery vividness also plays a decisive role in the effectiveness. In this study, the investigators developed a video game in which immune cells fight breast cancer cells, and through this video game, patients will be able to easily, actively, and vividly visualize their immune cells destroying the cancer. In the meantime, instead of being stressed, the patients will be playing games and having fun with imagery. Thus, the investigators developed a unique guided imagery complementary therapy called video-immunotherapy in the treatment of breast cancer. It is predicted that the immune system of the person playing the video game would be stimulated to exert an anti-tumoral effect. In this study, breast cancer patients will play the video immunotherapy or a control placebo video game in addition to their current treatment (neoadjuvant chemotherapy). The effect of the video immunotherapy on the course of the disease, physiological symptoms, and psychological well-being of the patients will be measured, and the effect of the game on the immune cells of the patients will be analyzed in detail.

ELIGIBILITY:
Inclusion Criteria:

* having locally advanced breast cancer
* To be over 18 years old
* Volunteering to participate in the study
* ECOG performance score of 0-1
* To be able to communicate in Turkish
* Obtaining written informed consent for participation in the study

Exclusion Criteria:

* History of epilepsy and similar seizures
* History of cognitive impairment such as dementia, Alzheimer's disease
* Major depression or suicidal tendencies
* Traumatic brain injury
* Lack of sight, hearing or use of hands
* Previous history of cancer other than breast cancer
* Chronic use of immunosuppressive drugs (e.g. steroids)
* Active immunodeficiency
* Having any disability to play video games

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only cisgender women
Enrollment: 80 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Depression Anxiety Stress Scale (DASS-42) total score | Experimental and control group patients will answer questionnaires to monitor their psychological status and physiological symptoms 3 times in total: baseline (month 0), during the treatment (month 3) and at the end of treatment (month 5-6).
  The Depression Anxiety Stress Scale (DASS-42) is a self-reported questionnaire designed to measure negative emotional states across three subscales: depression, anxiety, and stress. The total score is calculated by summing all 42 items.
  Minimum value: 0 Maximum value: 126 (42 items × 0-3 Likert scale)
  Score interpretation: Higher scores indicate worse psychological distress.
Change from baseline in Edmonton Symptom Assessment System-revised (ESAS-r) total symptom score | Baseline (Month 0), during treatment (Month 3), and end of treatment (Month 5-6)
  The Edmonton Symptom Assessment System-revised (ESAS-r) is a patient-reported outcome measure assessing the severity of common cancer-related symptoms, including pain, fatigue, nausea, depression, anxiety, drowsiness, appetite, well-being, shortness of breath, and an optional additional symptom. Each symptom is rated on a numeric scale.
  Minimum value: 0 Maximum value: 100 (10 symptoms × 0-10 numeric rating scale)
  Score interpretation: Higher scores indicate worse symptom burden.
Change from baseline in frequency of immune cell subsets in peripheral blood and tumor tissue | Peripheral blood: Baseline (Month 0) and end of treatment (Month 5-6) Tumor tissue: End of treatment (Month 5-6)
  The frequency of immune cell subsets involved in breast cancer immunity will be assessed by flow cytometry. The analyzed cell populations include CD4⁺ T cells, CD8⁺ T cells, regulatory T cells (Treg), NK cells, monocytes in peripheral blood and tumor tissue, and myeloid-derived suppressor cells, as well as M1 and M2 macrophages in tumor tissue only. Cell frequencies will be reported as a percentage of CD45⁺ live cells.
  Unit of Measure: Percentage (%)
Change from baseline in activation marker expression on immune cell subsets | Peripheral blood: Baseline (Month 0) and end of treatment (Month 5-6) Tumor tissue: End of treatment (Month 5-6)
  Activation status of immune cells will be evaluated by flow cytometry based on the expression of activation markers. NK cells and T cell subsets will be assessed using CD25, CD69, and HLADR expression, while monocytes and macrophages will be assessed using CD86 and HLADR expression. Activation will be reported as median fluorescence intensity (MFI).
  Unit of Measure: Median fluorescence intensity (MFI)
Change from baseline in tumor size measured by ultrasound and mammography for the assessment of the effects on disease progression | Baseline (Month 0), mid-treatment (Month 3), and end of treatment (Month 5-6)
  Tumor size will be assessed using standard clinical imaging methods, including ultrasound and mammography, to evaluate disease progression in patients receiving the UMAY video-immunotherapy or placebo control intervention.
  Tumor size will be recorded as the largest tumor diameter (in millimeters), according to routine clinical assessment.
  Unit of Measure: Millimeters (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Sag, Ph.D., Principal Investigator — Izmir Biomedicine and Genome Center
Locations (3):
- Turkey (Türkiye) (3):
  - Dokuz Eylul University Hospital, Izmir, Balcova
  - Akdeniz University Hospital, Antalya, Konyaaltı
  - Antalya Training and Research Hospital, Antalya, Muratpasa

IPD SHARING:
Plan to Share IPD: Yes
We plan to share de-identified IPD through controlled access after publication. Shared variables will include DASS and ESAS scores at baseline, mid-treatment and end-of-treatment; tumor size by ultrasound/mammography at the same time points; and flow-cytometry profiles of CD4+, CD8+, Treg, NK cells, monocytic cells from blood (baseline and month 5-6) and tumor tissue (month 5-6). All data will be anonymized and no direct identifiers will be released. Access will require ethics approval and a data-use agreement. Access will be prioritized for investigators conducting non-commercial research aimed at advancing breast-cancer immunotherapy or improving statistical/clinical reproducibility.
Supporting Information: Study Protocol, CSR
Time Frame: Data will be shared upon reasonable request following publication of primary results, conditional on ethics approval and data-use agreement outlining scientific purpose and confidentiality obligations.
Access Criteria: investigators conducting non-commercial research